CLINICAL TRIAL: NCT00013481
Title: Coordination of Hemiparetic Movement After Post-Stroke Rehabilitation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Duncan, Pamela - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2116
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2009-11-10 (Estimated); Status verified 2009-11

CONDITIONS: Stroke
Keywords: stroke, hemiparesis, CNS, motor coordination
MeSH Terms: conditions — Stroke; Paresis | interventions — Stroke Rehabilitation

ARMS (1):
- 1 (Other)
  Interventions: Procedure: Stroke Rehabilitation

INTERVENTIONS:
Procedure: Stroke Rehabilitation

SUMMARY:
This study will determine whether a therapeutic exercise program for improving motor coordination in locomotor tasks in post-stroke, hemiparesis patients will result in CNS recovery. The study will develop relationships between the improved motor performance and motor coordination during the locomotor task and the functional effects of the exercise program(e.g., gait variables.)

DETAILED DESCRIPTION:
Primary objective of this study is to determine whether a therapeutic exercise program which targets the functional recovery of persons with the post-stroke hemiparesis results in CNS recovery (improved motor coordination). They will determine whether motor coordination during a locomotor task is improved after an exercise program. They will then develop relationships between the improved motor performance and motor coordination during the locomotor task and the functional effects of the exercise program(e.g., gait variables) Overall goal is to develop a more rational basis for the design of stroke rehabilitation programs which target individuals most likely to recover and which are based on physiological principles. This study will supplement an NIH funded randomized clinical trial to evaluate a post-stroke exercise program designed to increase balance, strength, and endurance. Study will include 60-70 prospective patients enrolled in the randomized clinical trial at Kansas University Center on Aging. between Oct 1999 and Oct 2001.

ELIGIBILITY:
Inclusion Criteria:

Functionally impaired elderly

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2000-01; Primary Completion 2003-09 (Actual); Study Completion 2003-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela W. Duncan, PhD MA BS, Principal Investigator — North Florida/South Georgia Veterans Health System
Locations (1):
- North Florida/South Georgia Veterans Health System, Gainesville, Florida, United States